CLINICAL TRIAL: NCT00985426
Title: An Observer-Blinded, Randomized Study Comparing the Safety and Immunogenicity of HEPLISAV-B® to Licensed Vaccine (Engerix-B®) Among Adults(18 to 75 Years of Age) With Chronic Kidney Disease (CKD)
Brief Title: Comparing Safety and Immunogenicity of HEPLISAV-B® to Engerix-B® in Chronic Kidney Disease (CKD) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DV2-HBV-17; 2009-015877-11 (EudraCT Number)
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; kidney failure; kidney failure,chronic; chronic kidney failure; hepatitis B virus (HBV) vaccine; hepatitis B vaccine; hepatitis B; hepatitis; HBV; prevention and control; dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Kidney Failure, Chronic; Hepatitis B; Hepatitis | interventions — Heplisav-B; Hepatitis B Vaccines; Engerix-B; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HEPLISAV-B (Experimental): 0.5 mL HEPLISAV-B and 0.5 mL Placebo
  Interventions: Biological: HEPLISAV-B; Other: Placebo
- Engerix-B (Active Comparator): 2.0 mL Engerix-B
  Interventions: Biological: Engerix-B

INTERVENTIONS:
Biological: HEPLISAV-B — Intramuscular (IM) injections of HEPLISAV-B at Weeks 0, 4, and 24
  Other Names: Hepatitis B vaccine (recombinant), adjuvanted
  Arms: HEPLISAV-B
Biological: Engerix-B — Intramuscular (IM) injections at Weeks 0, 4, 8, and 24
  Other Names: Hepatitis B vaccine (recombinant)
  Arms: Engerix-B
Other: Placebo — Placebo(saline) intramuscular (IM) injection at Week 8
  Other Names: Saline
  Arms: HEPLISAV-B

SUMMARY:
The purpose of the study is to demonstrate the safety and immunogenicity of a new investigational hepatitis B virus vaccine, HEPLISAV-B, in patients 18 to 75 years of age who have progressive loss of kidney function.

ELIGIBILITY:
Inclusion Criteria:

* be 18 to 75 years of age;
* progressive loss of renal function as defined by glomerular filtration rate (GFR) ≤ 45 mL/min/1.73 m²;
* be clinically stable in the opinion of the investigator;
* be serum negative for HBsAg, anti-HBsAg, antibody to hepatitis B core antigen (HBcAg), Hepatitis C virus (HCV), and human immunodeficiency virus (HIV);
* if a woman of childbearing potential, agree to consistently use a highly effective method of birth control from screening visit through the treatment phase and for up to 28 days after the last injection;
* is not scheduled to undergo a kidney transplant in the next 12 months;
* be able and willing to provide informed consent.

Exclusion Criteria:

* if female, is pregnant, breastfeeding, or planning a pregnancy;
* has a history of or is considered by the investigator to be at high risk for recent exposure to HBV, HCV, or HIV; for example, current intravenous drug use, has unprotected sex with known HBV/HIV positive partner;
* has known history of autoimmune disease;
* has previously received any HBV vaccine;
* has a history of sensitivity to any component of study vaccines;
* has current illness other than renal disease or has substance or alcohol abuse that in the opinion of the investigator would interfere with compliance or with interpretation of the study results;
* is undergoing chemotherapy or expected to receive chemotherapy during the study period; has a diagnosis of cancer within the last 5 years other than squamous or basal cell carcinoma of the skin;
* has uncontrolled diabetes or hypertension;
* is unwilling or unable to comply with all the requirements of the protocol;
* has received any blood products or immunoglobulin within 3 months prior to study entry, or likely to require infusion of blood products during the study period;
* has received the following prior to the first injection:
* 3 days: erythropoietin (exclusionary window does not apply for subjects on dialysis)
* 7 days: intravenous iron
* 21 days: any inactivated virus vaccine
* 28 days:
* any live virus vaccine
* systemic corticosteroids (more than 3 consecutive days) or other immunomodulators or immune suppressive medication, with the exception of inhaled steroids
* granulocyte or granulocyte-macrophage colony-simulating factor (G/GM-CSF), any other investigational medicinal agent
* At any time: an injection of deoxyribonucleic acid plasmids or oligonucleotide

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Janssen, MD, Study Director — Dynavax Technologies Corporation
Locations (1):
- Clinical Research Associates of Tidewater, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Janssen RS, Mangoo-Karim R, Pergola PE, Girndt M, Namini H, Rahman S, Bennett SR, Heyward WL, Martin JT. Immunogenicity and safety of an investigational hepatitis B vaccine with a toll-like receptor 9 agonist adjuvant (HBsAg-1018) compared with a licensed hepatitis B vaccine in patients with chronic kidney disease. Vaccine. 2013 Nov 4;31(46):5306-13. doi: 10.1016/j.vaccine.2013.05.067. Epub 2013 May 30. PMID 23727422
- See also: Related Info — http://www.dynavax.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- HEPLISAV-B: To mimic the Engerix dosing regimen and to maintain the blind, subjects randomized to the HEPLISAV group received 0.5 mL HEPLISAV and 0.5 mL Placebo (saline) via intramuscular (IM) injections at Weeks 0, 4, and 24.
  To mimic the Engerix dosing regimen and to maintain the blind, subjects also received two 0.5-mL IM injections of Placebo (saline) at Week 8.
- Engerix-B: Subjects randomized to the Engerix-B group received two 1.0-mL IM injections of Engerix-B at Weeks 0, 4, 8, and 24.
Period: Overall Study
Arm/Group | HEPLISAV-B | Engerix-B
Started | 258 | 263
Completed | 215 | 219
Not Completed | 43 | 44
Not completed — Adverse Event | 0 | 1
Not completed — Subject Non-Compliance | 3 | 3
Not completed — Withdrawal by Subject | 12 | 16
Not completed — Lost to Follow-up | 8 | 10
Not completed — Death | 7 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Lack of seroprotection at protocol-specified timepoints | 11 | 11

BASELINE CHARACTERISTICS:
Population: Safety population includes randomized participants who received at least 1 study injection.
Groups:
- HEPLISAV-B: Participants randomized to the HEPLISAV-B group received 0.5 mL HEPLISAV-B and 0.5 mL Placebo (saline) via intramuscular (IM) injections at Weeks 0, 4, and 24.
  Participants also received two 0.5-mL IM injections of Placebo (saline) at Week 8.
- Engerix-B: Participants randomized to the Engerix-B group received two 1.0-mL IM injections of Engerix-B at Weeks 0, 4, 8, and 24.
- Total: Total of all reporting groups
Arm/Group | HEPLISAV-B | Engerix-B | Total
Number analyzed (Participants) | 254 | 262 | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (9.1) | 61.3 (9.7) | 61.3 (9.4)
Age, Customized [Count of Participants; unit: Participants]
  Age Strata: 18 to 39 years | 3 | 11 | 14
  Age Strata: 40 to 55 years | 58 | 52 | 110
  Age Strata: 56 to 75 years | 193 | 199 | 392
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 104 | 198
  Male | 160 | 158 | 318
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65 | 71 | 136
  Not Hispanic or Latino | 189 | 191 | 380
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 44 | 47 | 91
  White | 204 | 203 | 407
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 34.05 (8.45) | 32.15 (6.94) | 33.09 (7.77)
Smoking status [Count of Participants; unit: Participants]
  Yes | 34 | 43 | 77
  No | 220 | 219 | 439
Glomerular Filtration Rate (GFR) at Screening [Count of Participants; unit: Participants]
  GFR ≤ 15 mL/min/1.73 m2 | 39 | 55 | 94
  GFR 16 - 30 mL/min/1.73 m2 | 99 | 96 | 195
  GFR ≥ 31 mL/min/1.73 m2 | 116 | 111 | 227
Screening Creatinine [Mean (Standard Deviation); unit: mg/dL] | 2.66 (1.42) | 2.82 (1.64) | 2.74 (1.53)
History of Type 2 Diabetes Mellitus [Count of Participants; unit: Participants] | 173 | 161 | 334

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection Rate (SPR) = Percentage of Participants Who Have a Seroprotective Immune Response
Description: SPR is the percentage of participants who have a seroprotective immune response (antibody level to anti-HBsAg greater than or equal to 10 milli-international unit [mIU]/mL) after HEPLISAV-B compared to that after Engerix-B.
Time Frame: Week 28
Population: Modified Intent-to-Treat (mITT) population comprises all randomized participants who received at least 1 study injection and had at least 1 post-injection immunogenicity evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | HEPLISAV-B | Engerix-B
Number analyzed (Participants) | 227 | 242
Participants | 204 | 198
Statistical Analysis 1: Comparison: HEPLISAV-B vs Engerix-B; Two-sided 95% confidence intervals (CIs) of the difference in seroprotection rates (SPR) between the HEPLISAV-B group and the Engerix-B group at 28 weeks was computed using the Newcombe score method with continuity correction; Test type: Non-Inferiority — Non-inferiority is achieved if the lower limit of the two-sided 95% CI was greater than -10%; SPR Difference (%) = 8, 95% CI 2-sided [1.7 to 14.3] — SPR difference = SPR for HEPLISAV-B minus SPR for Engerix-B
Statistical Analysis 2: Comparison: HEPLISAV-B vs Engerix-B; Two-sided 95% CIs of the difference in SPR between the HEPLISAV-B group and the Engerix-B group at 28 weeks was computed using the Newcombe score method with continuity correction; Test type: Superiority — Superiority is achieved if the lower limit of the two-sided 95% CI was greater than 0%; SPR Difference (%) = 8, 95% CI 2-sided [1.7 to 14.3]

2. Secondary Outcome: Reactogenicity as Measured by the Percentage of Participants With Local and Systemic Post-injection Reactions Within 7 Days After Each Injection Visit
Description: Local reactions include redness greater than or equal to 25 mm, swelling greater than or equal to 25 mm, and pain.
  Systemic reactions include malaise, headache, myalgia, fatigue, and fever (temperature greater than or equal to 38ºC).
  This table presents post-injection reactions at active injection visits only. Post-injection reactions after the third (placebo) injection visit in the HEPLISAV-B group are not included.
Time Frame: 7 days after each injection visit (Weeks 0, 4, 8, and 24)
Population: Safety population includes randomized participants who received at least 1 study injection.
Measure: Count of Participants; unit: Participants
Arm/Group | HEPLISAV-B | Engerix-B
Number analyzed (Participants) | 254 | 262
Participants
  Local reactions | 73 | 90
  Systemic reactions | 85 | 91

3. Secondary Outcome: Seroprotection Rate (SPR) = Percentage of Participants Who Have a Seroprotective Immune Response at Weeks 4, 8, 12, 18, 24, 28, 36, 44, and 52
Description: as for outcome 1
Time Frame: Weeks 4, 8, 12, 18, 24, 28, 36, 44, and 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants (SPR)
Arm/Group | HEPLISAV-B | Engerix-B
Number analyzed (Participants) | 247 | 260
percentage of participants (SPR)
  Week 4: number analyzed (Participants) | 247 | 258
  Week 4 | 5.7 [3.1 to 9.3] | 6.2 [3.6 to 9.9]
  Week 8: number analyzed (Participants) | 241 | 257
  Week 8 | 48.1 [41.7 to 54.6] | 20.2 [15.5 to 25.7]
  Week 12: number analyzed (Participants) | 238 | 248
  Week 12 | 65.1 [58.7 to 71.2] | 50.8 [44.4 to 57.2]
  Week 18: number analyzed (Participants) | 236 | 247
  Week 18 | 73.7 [67.6 to 79.2] | 59.5 [53.1 to 65.7]
  Week 24: number analyzed (Participants) | 235 | 246
  Week 24 | 78.7 [72.9 to 83.8] | 62.2 [55.8 to 68.3]
  Week 28: number analyzed (Participants) | 227 | 242
  Week 28 | 89.9 [85.2 to 93.5] | 81.8 [76.4 to 86.5]
  Week 36: number analyzed (Participants) | 222 | 234
  Week 36 | 86.9 [81.8 to 91.1] | 80.3 [74.7 to 85.2]
  Week 44: number analyzed (Participants) | 218 | 220
  Week 44 | 83.9 [78.4 to 88.6] | 78.6 [72.6 to 83.9]
  Week 52: number analyzed (Participants) | 217 | 220
  Week 52 | 84.3 [78.8 to 88.9] | 77.3 [71.2 to 82.6]

4. Secondary Outcome: Percentage of Participants With Anti-HBsAg Greater Than or Equal to 100 mIU/mL at Weeks 4, 8, 12, 18, 24, 28, 36, 44, and 52
Time Frame: Weeks 4, 8, 12, 18, 24, 28, 36, 44, and 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % participants
Arm/Group | HEPLISAV-B | Engerix-B
Number analyzed (Participants) | 247 | 260
% participants
  Week 4: number analyzed (Participants) | 247 | 258
  Week 4 | 3.6 [1.7 to 6.8] | 2.7 [1.1 to 5.5]
  Week 8: number analyzed (Participants) | 241 | 257
  Week 8 | 19.5 [14.7 to 25.1] | 7 [4.2 to 10.8]
  Week 12: number analyzed (Participants) | 238 | 248
  Week 12 | 27.3 [21.8 to 33.4] | 22.2 [17.2 to 27.9]
  Week 18: number analyzed (Participants) | 236 | 247
  Week 18 | 38.6 [32.3 to 45.1] | 25.9 [20.6 to 31.8]
  Week 24: number analyzed (Participants) | 235 | 246
  Week 24 | 45.1 [38.6 to 51.7] | 28.5 [22.9 to 34.5]
  Week 28: number analyzed (Participants) | 227 | 242
  Week 28 | 73.6 [67.3 to 79.2] | 63.2 [56.8 to 69.3]
  Week 36: number analyzed (Participants) | 222 | 234
  Week 36 | 68.9 [62.4 to 74.9] | 59 [52.4 to 65.3]
  Week 44: number analyzed (Participants) | 218 | 220
  Week 44 | 67.9 [61.3 to 74] | 54.5 [47.7 to 61.3]
  Week 52: number analyzed (Participants) | 217 | 220
  Week 52 | 66.8 [60.1 to 73] | 49.1 [42.3 to 55.9]

5. Secondary Outcome: Serum Anti-HBsAg Geometric Mean Concentration (GMC) at Weeks 4, 8, 12, 18, 24, 28, 36, 44, and 52
Time Frame: Weeks 4, 8, 12, 18, 24, 28, 36, 44, and 52
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HEPLISAV-B | Engerix-B
Number analyzed (Participants) | 247 | 260
mIU/mL
  Week 4: number analyzed (Participants) | 247 | 258
  Week 4 | .4 [.3 to .5] | .3 [.2 to .3]
  Week 8: number analyzed (Participants) | 241 | 257
  Week 8 | 8.1 [5.6 to 11.7] | .9 [.7 to 1.3]
  Week 12: number analyzed (Participants) | 238 | 248
  Week 12 | 16.5 [11.7 to 23.4] | 7.2 [5 to 10.4]
  Week 18: number analyzed (Participants) | 236 | 247
  Week 18 | 33 [23.4 to 46.6] | 12 [8.4 to 17.2]
  Week 24: number analyzed (Participants) | 235 | 246
  Week 24 | 44.3 [31.6 to 62.3] | 15.1 [10.6 to 21.5]
  Week 28: number analyzed (Participants) | 227 | 242
  Week 28 | 587.1 [386.7 to 891.4] | 156.5 [103.6 to 236.3]
  Week 36: number analyzed (Participants) | 222 | 234
  Week 36 | 302.3 [200.5 to 456] | 104.2 [69.8 to 155.6]
  Week 44: number analyzed (Participants) | 218 | 220
  Week 44 | 214.5 [145.2 to 316.8] | 71.2 [48.1 to 105.5]
  Week 52: number analyzed (Participants) | 217 | 220
  Week 52 | 170.8 [117 to 249.2] | 51 [34.7 to 74.9]

6. Secondary Outcome: SPR of Participants With Type 2 Diabetes Mellitus at Week 28
Description: as for outcome 1
Time Frame: Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HEPLISAV-B | Engerix-B
Number analyzed (Participants) | 153 | 150
Participants | 137 | 115
Statistical Analysis 1: Comparison: HEPLISAV-B vs Engerix-B; Two-sided 95% CIs of the difference in SPRs between the HEPLISAV group and the Engerix-B group at 28 weeks was computed using the Newcombe score method with continuity correction; Test type: Superiority — Superiority is achieved if the lower limit of the two-sided 95% CI was greater than 0%; SPR Difference (%) = 12.9, 95% CI 2-sided [4.4 to 21.2]

ADVERSE EVENTS:
Time Frame: Reporting period for adverse events (AEs) that were not serious adverse events (SAEs) was the time from the first study injection until Week 28. Reporting period for SAEs was the time from the signing of the informed consent form until Week 52 (or completion of the participant's participation in the study).
Arm/Group | HEPLISAV-B | Engerix-B
All-Cause Mortality (participants affected / at risk) | 7/254 | 3/262
Serious Adverse Events (participants affected / at risk) | 68/254 | 76/262
Other Adverse Events (participants affected / at risk) | 140/254 | 146/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV-B (N=254) | Engerix-B (N=262)
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 2
Angina pectoris (Cardiac disorders) | 0 | 3
Angina unstable (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 8 | 8
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 5
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enlarged uvula (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 1
Hernia obstructive (General disorders) | 1 | 0
Medical device complication (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 3
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Fungal peritonitis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 2
Perineal abscess (Infections and infestations) | 0 | 1
Pneumococcal bacteraemia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 4
Pneumonia escherichia (Infections and infestations) | 1 | 0
Renal cyst infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 2 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 3 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Azotaemia (Renal and urinary disorders) | 0 | 3
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal cyst ruptured (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 5 | 7
Renal failure chronic (Renal and urinary disorders) | 9 | 12
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 3
Victim of homicide (Social circumstances) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 4
Hypertensive crisis (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 2
Malignant hypertension (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 2
Steal syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HEPLISAV-B (N=254) | Engerix-B (N=262)
Anaemia (Blood and lymphatic system disorders) | 9 | 11
Cataract (Eye disorders) | 7 | 3
Constipation (Gastrointestinal disorders) | 11 | 11
Diarrhoea (Gastrointestinal disorders) | 11 | 10
Nausea (Gastrointestinal disorders) | 11 | 13
Vomiting (Gastrointestinal disorders) | 6 | 8
Fatigue (General disorders) | 16 | 13
Oedema peripheral (General disorders) | 16 | 13
Bronchitis (Infections and infestations) | 9 | 8
Gastroenteritis (Infections and infestations) | 7 | 2
Nasopharyngitis (Infections and infestations) | 13 | 18
Sinusitis (Infections and infestations) | 7 | 7
Upper respiratory tract infection (Infections and infestations) | 11 | 11
Urinary tract infection (Infections and infestations) | 12 | 7
Blood creatine phosphokinase increased (Investigations) | 7 | 5
Gout (Metabolism and nutrition disorders) | 7 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 11 | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 4 | 8
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 11
Dizziness (Nervous system disorders) | 4 | 8
Headache (Nervous system disorders) | 9 | 8
Insomnia (Psychiatric disorders) | 6 | 1
Renal failure chronic (Renal and urinary disorders) | 11 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 8
Hypertension (Vascular disorders) | 8 | 18
Hypotension (Vascular disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less